CLINICAL TRIAL: NCT01869075
Title: Toronto Thromboprophylaxis Patient Safety Initiative (TOPPS): A Cluster Randomized Trial
Brief Title: Toronto Thromboprophylaxis Patient Safety Initiative
Acronym: TOPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: North York General Hospital (Other); Michael Garron Hospital (Other); Trillium Health Centre (Other); Lakeridge Health Corporation (Other); York Central Hospital, Ontario (Other); Scarborough General Hospital (Other); Markham Stouffville Hospital (Other)
Responsible Party: Principal Investigator, Artemis Diamantouros, KT Pharmacist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 019-2006
Record Dates: First submitted 2013-04-03; First posted 2013-06-05 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Venous Thromboembolism
Keywords: Quality Improvement; Patient Safety; Knowledge Translation
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- AMI - Knowledge Translation toolkit (Experimental): AMI - Knowledge Translation (KT) toolkit includes use of pre-printed orders, audit and feedback, pharmacist as a reminder and education of staff
  Interventions: Other: Knowledge Translation (KT) toolkit
- AMI - Usual Care (No Intervention): Usual care
- MGS - Knowledge Translation Toolkit (Experimental): Knowledge Translation toolkit involves use of pre-printed orders, audit and feedback, pharmacist as reminder and education of staff
  Interventions: Other: Knowledge Translation (KT) toolkit
- MGS - Usual Care (No Intervention): Usual Care
- HFS - Knowledge Translation Toolkit (Experimental): Knowledge Translation Toolkit consists of pre-printed orders, audit and feedback, pharmacist as a reminder and education of staff
  Interventions: Other: Knowledge Translation (KT) toolkit
- HFS - Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Knowledge Translation (KT) toolkit — KT toolkit consists of: use of pre-printed orders, use of pharmacist as project lead and human reminder for prescribing, audit and feedback, education for staff
  Other Names: AMI - Knowledge Translation (KT) toolkit; MGS - Knowledge Translation (KT) toolkit; HFS - Knowledge Translation (KT) toolkit
  Arms: AMI - Knowledge Translation toolkit; HFS - Knowledge Translation Toolkit; MGS - Knowledge Translation Toolkit

SUMMARY:
Venous thromboembolism (VTE), which includes deep vein thrombosis (DVT) and pulmonary embolism (PE, is one of the common and preventable complications of hospital stay. VTE prophylaxis through the use of evidence-based anticoagulant medication options or mechanical prophylaxis have been shown to reduce this risk and improve patient safety. Despite an abundance of evidence, use of VTE prophylaxis remains low.

This study assesses the effectiveness of quality improvement strategies (use of pre-printed orders, audit and feedback, involvement of the pharmacist as project need and as a reminder to the physician, and education of staff) on use of appropriate VTE prophylaxis. The study aims to measure if the use of these strategies improves the use of VTE prophylaxis and therefore, improves patient safety and patient care by reducing the risk of developing DVT or PE.

DETAILED DESCRIPTION:
The study includes 8 Toronto area hospitals consisting of 7 community hospital and one academic health sciences centre.

Three patient groups at each site are included in the study: patients admitted for: Acute Medical Illness (AMI), Major General Surgery (MGS) and Hip Fracture Surgery (HFS). Patients had to be at least 18 years old and be considered at risk for VTE according to the American College of Chest Physicians (CHEST) guidelines.

The study design is a cluster randomized trial where each patient group at each site is a cluster.

A baseline chart audit of approximately 50 patients in each group at each site was conducted to determine an intraclass coefficient and proportion of adherence.

The main outcome measure was the rate of prescribing appropriate prophylaxis in patients at risk. This was calculated as the number of at risk patients receiving appropriate prophylaxis / the number of at risk patients for whom prophylaxis is indicated.

Based on the baseline results, it was estimated that a sample size of 432 would be needed for the intervention phases. A sample of 720 patients (15 in each cluster at each site) was included.

The study is broken down into three phases: baseline, phase 1 and phase 2. At baseline, all groups received usual care. At phase 1, one cluster at each site was randomized to intervention while the other two served as control. In phase 2, 2 groups received intervention while one continued to serve as control. Each of the phases, phase 1 and 2 had 360 unique patients. Patients in baseline were not included in phase 1 or 2 and patients in phase 1 were not included in phase 2.

The main outcome measure was prescribing of appropriate VTE prophylaxis. A chart audit was used to collect data at baseline, end of phase 1 and end of phase 2.

Each phase is approximately 1 year in length. Analysis involves descriptive statistics using counts and proportions to capture rates of appropriate VTE prophylaxis and rates of non-adherence. A logistic regression model will be used to compare rates of appropriate VTE prophylaxis over time within groups adjusted for clustering.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* at risk for VTE

Exclusion Criteria:

* on therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1895 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Geerts, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of study sites not individual patients.
Pre-assignment Details: After site enrolment, baseline data was collected for all sites in order to establish sample size for phases 1 and 2.
Groups:
- AMI - Usual Care; MGS - Usual Care; HFS - Usual Care: Usual care provided at the hospital
Period: Phase 0 (Baseline)
Arm/Group | AMI - Knowledge Translation Toolkit | AMI - Usual Care | MGS - Knowledge Translation Toolkit | MGS - Usual Care | HFS - Knowledge Translation Toolkit | HFS - Usual Care
Started | 0 (Phase 0 was the baseline phase. No intervention had been started.) | 418 | 0 (Phase 0 was the baseline phase. No intervention had been started.) | 416 | 0 (Phase 0 was the baseline phase. No intervention had been started.) | 341
Completed | 0 | 418 | 0 | 416 | 0 | 341
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1
Arm/Group | AMI - Knowledge Translation Toolkit | AMI - Usual Care | MGS - Knowledge Translation Toolkit | MGS - Usual Care | HFS - Knowledge Translation Toolkit | HFS - Usual Care
Started | 45 (Each phase of the study collected data on a unique set of patients.) | 75 (Each phase of the study collected data on a unique set of patients.) | 45 (Each phase of the study collected data on a unique set of patients.) | 75 (Each phase of the study collected data on a unique set of patients.) | 30 (Each phase of the study collected data on a unique set of patients.) | 90 (Each phase of the study collected data on a unique set of patients.)
Completed | 45 | 75 | 45 | 75 | 30 | 90
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | AMI - Knowledge Translation Toolkit | AMI - Usual Care | MGS - Knowledge Translation Toolkit | MGS - Usual Care | HFS - Knowledge Translation Toolkit | HFS - Usual Care
Started | 90 (Participants included in phase 2 of the study were not enrolled in phase 1. Each is a unique phase.) | 30 (Participants included in phase 2 of the study were not enrolled in phase 1. Each is a unique phase.) | 75 (Participants included in phase 2 of the study were not enrolled in phase 1. Each is a unique phase.) | 45 (Participants included in phase 2 of the study were not enrolled in phase 1. Each is a unique phase.) | 75 (Participants included in phase 2 of the study were not enrolled in phase 1. Each is a unique phase.) | 45 (Participants included in phase 2 of the study were not enrolled in phase 1. Each is a unique phase.)
Completed | 90 | 30 | 75 | 45 | 75 | 45
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data collection was conducted to establish baseline rates of appropriate prophylaxis. Baseline patients were not included in the active phases of the study.
Groups:
- AMI - Usual Care; MGS - Usual Care; HFS - Usual Care: Usual care as provided at the hospital.
- Total: Total of all reporting groups
Arm/Group | AMI - Knowledge Translation Toolkit | AMI - Usual Care | MGS - Knowledge Translation Toolkit | MGS - Usual Care | HFS - Knowledge Translation Toolkit | HFS - Usual Care | Total
Number analyzed (Participants) | 0 | 341 | 0 | 416 | 0 | 418 | 1175
Age, Customized [Number; unit: participants]
  18 years and older |  | 341 |  | 416 |  | 418 | 1175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | NA — Gender of participants was not collected |  | NA — Gender of participants was not collected |  | NA — Gender of participants was not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male |  | NA — Gender of participants was not collected |  | NA — Gender of participants was not collected |  | NA — Gender of participants was not collected | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Prescribed Appropriate VTE Prophylaxis
Description: Rates of appropriate VTE prophylaxis were determined as the number of patients who received VTE prophylaxis as a proportion of the number of patient at risk.
  Rates reported are for the active phases (phase 1 and phase 2) and compare intervention to control.
  Appropriate VTE prophylaxis was defined as:
  in "Hip Fracture Surgery" - evidence-based VTE prophylaxis ordered within 24 of admission, restarted within 24 hours after surgery and continued for at least 10 days post-discharge in "Major General Surgery" - evidence-based VTE prophylaxis ordered within 24 hours post-surgery and continued for the duration of hospital stay in "Acute Medical Illness" - evidence-based VTE prophylaxis ordered within 24 hours of admission and continued for the duration of hospital stay.
  Evidence-based VTE prophylaxis was determined to be according to the American College of Chest Physicians (ACCP) guidelines. The 9th version was the most current version at the time of the study.
Time Frame: End of study (end of phase 2) - measured over duration of hospital stay.
Population: The number of participants in the analysis was 720. In phase 1, there were 360 patients included and in phase 2, an additional 360 patients were included. The outcomes by end of study (end of phase 2) are reported. The patients in control (usual care) and intervention (Knowledge Translation toolkit) were compared.
Measure: Number; unit: percentage of patients
Arm/Group | AMI - Knowledge Translation Toolkit | AMI - Usual Care | MGS - Knowledge Translation Toolkit | MGS - Usual Care | HFS - Knowledge Translation Toolkit | HFS - Usual Care
Number analyzed (Participants) | 135 | 105 | 120 | 120 | 105 | 135
percentage of patients | 64 [0.89 to 3.36] | 62 [lower limit 0.89] | 67 | 54 | 85 | 76

ADVERSE EVENTS:
Time Frame: At one point in time at phase 1 and phase 2. Phase 1 and 2 were approx 1 year apart. Adverse events were only captured if they occured in the participants in the audit sample during their hospital admission.
Arm/Group | AMI - Knowledge Translation Toolkit | AMI - Usual Care | MGS - Knowledge Translation Toolkit | MGS - Usual Care | HFS - Knowledge Translation Toolkit | HFS - Usual Care
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/105 | 0/120 | 0/120 | 0/105 | 0/135
Other Adverse Events (participants affected / at risk) | 0/135 | 0/105 | 0/120 | 0/120 | 0/105 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No